CLINICAL TRIAL: NCT07231770
Title: A Controlled Study on the Prophylaxis of Pneumocystis Jirovecii Pneumonia With Fixed-dose Compound Sulfamethoxazole Tablets of Different Maintenance Durations After Renal Transplantation
Brief Title: Sulfamethoxazole Prophylaxis Duration After Renal Transplantation
Acronym: SPDART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USTC-PJP-Pro; 2023-ky041 (Other: The First Affiliated Hospital of University of Science and Technology of China (USTC))
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Fever; Chest Tightness
MeSH Terms: conditions — Fever

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A group (Other): 6-month SMZ prophylaxis
  Interventions: Other: Time-driven dosing
- B group (Other): 12-month SMZ prophylaxis
  Interventions: Other: Time-driven dosing
- C group (Other): 18-month SMZ prophylaxis
  Interventions: Other: Time-driven dosing

INTERVENTIONS:
Other: Time-driven dosing — The total sample size required for the study is 450 cases. Patients will then be screened for enrollment according to the inclusion and exclusion criteria, and randomly assigned to Groups A, B, and C in a 1:1:1 ratio, with 150 patients in each group. Group A will receive TMP-SMX prophylaxis against PJP for 6 months, while Groups B and C will each receive TMP-SMX prophylaxis against PJP for 12 months.

SUMMARY:
Renal transplantation is the most ideal and effective treatment for end-stage renal disease. Pneumocystis jirovecii pneumonia (PJP) is one of the most common pulmonary infections after renal transplantation, with high morbidity and mortality that seriously affects patients' prognosis and survival. PJP can be prevented with drugs, and trimethoprim-sulfamethoxazole (TMP-SMX) is the first-choice prophylactic agent. However, there is no clear definition of the prophylactic course of TMP-SMX in domestic and international guidelines. Most of the prophylactic durations for PJP are based on the clinical experience of physicians, ranging from 6 to 12 months across different transplant centers. Multiple studies have shown that some patients still develop PJP more than one year after renal transplantation. Previous research by our team found that PJP has a peak incidence around 9 months after renal transplantation, with a second peak occurring between 10 and 15 months. This study aims to adopt a single-center, randomized, parallel-controlled trial design, planning to enroll 450 patients after renal transplantation. It will investigate the impact of different prophylactic courses of TMP-SMX on the incidence of PJP, and explore whether long-term prophylaxis is more reasonable and effective than short-term prophylaxis. Meanwhile, during follow-up, the peak serum concentration of SMZ in patients will be measured to analyze the relationship between SMZ serum concentration and the occurrence of PJP as well as adverse reactions. A clinical prediction model will be constructed to reveal the effective concentration range of TMP-SMX for prophylactic use. This will further optimize the prophylactic regimen, provide practical guidance for clinical practice, reduce the morbidity and mortality of PJP, and improve prognosis.

ELIGIBILITY:
Diagnostic Criteria for PJP (meeting one of the following criteria is sufficient):

1. Detection of Pneumocystis jirovecii via sputum Gomori methenamine silver (GMS) stain.
2. According to guidelines/consensus: Positive direct immunofluorescence assay and/or positive polymerase chain reaction (PCR) assay on induced sputum or bronchoalveolar lavage fluid (BALF) specimens.
3. Detection of Pneumocystis jirovecii strains in sputum, blood, or bronchoalveolar lavage fluid (BALF) by metagenomic next-generation sequencing (mNGS).

Inclusion Criteria:

* Subjects must meet all the following conditions to be enrolled: (1) Age: 18-70 years old; (2) Post-renal transplantation; (3) Voluntarily participate in this clinical study, be able to cooperate with researchers to conduct the study, and sign the informed consent form.

Exclusion Criteria:

* Criteria: Subjects with any of the following conditions shall be excluded from the trial: (1) HIV-positive; (2) History of TMP-SMX allergy; (3) Glucose-6-phosphate dehydrogenase (G6PD) deficiency; (4) Megaloblastic anemia; (5) Multiorgan transplantation; (6) Complicated with tumor; (7) Complicated with connective tissue disease; (8) Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of PJP | 18 months after the end of treatment

SECONDARY OUTCOMES:
adverse reaction rate | 18 month

CONTACTS AND LOCATIONS:
Locations (1):
- No. 17, Lujiang Road, Luyang District, Hefei City, Anhui Province, China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No